CLINICAL TRIAL: NCT04506242
Title: Efficacy and Safety of Camrelizumab (SHR-1210) With Apatinib as Neoadjuvant Therapy for Participants With Resectable Non-Small Cell Lung Cancer: a Single-Arm, Phase II Study
Brief Title: Camrelizumab With Apatinib as Neoadjuvant Therapy for Participants With Resectable Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shugeng Gao, chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-II-006
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: NSCLC
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib+ Neoadjuvant/Adjuvant camrelizumab (Experimental): Neoadjuvant: Prior to surgery, participants receive 3 cycles (cycle length: 2 weeks) of camrelizumab [200 mg, intravenous (IV); given on cycle day 1] in combination with apatinib ,5 days on 2days off].
  Adjuvant: 4-8 weeks following surgery, participants receive up to 12 cycles (cycle length: 2 weeks) of camrelizumab [200 mg, IV; given on cycle day 1]. Participants who can not able to benefit from immunotherapy will not receive camrelizumab adjuvant therapy.
  Interventions: Drug: SHR-1210; Drug: Apatinib

INTERVENTIONS:
Drug: SHR-1210 — PD-1
  Other Names: camrelizumab
Drug: Apatinib — VEGFR2

SUMMARY:
This trial will evaluate the safety and efficacy of Camrelizumab (SHR-1210) in combination with apatinib neoadjuvant therapy before surgery [neoadjuvant phase], followed by camrelizumab alone after surgery [adjuvant phase] in participants with resectable stage IIA-IIIA, and resectable IIIB (T3N2) non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This trial will evaluate the safety and efficacy of camrelizumab in combination with apatinib neoadjuvant chemotherapy (NAC) before surgery [neoadjuvant phase], followed by camrelizumab alone after surgery [adjuvant phase] in participants with resectable stage II, IIIA, and resectable IIIB (T3N2) non-small cell lung cancer (NSCLC). The primary hypotheses of this study are that neoadjuvant camrelizumab in combination with apatinib, followed by surgery and adjuvant camrelizumab will improve: 1)MPR assessed by investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) ; 2) event free survival (EFS) and 3) overall survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 -70 years, male and female are not limited;
2. Patients with ECOG score of 0-1;
3. The thoracic surgeon judges the patients without contraindications;
4. Patients with early stage non-small cell lung cancer confirmed by histopathology; patients with stage iia-iiib non-small cell lung cancer (IIIB only limited to T3N2), which can be resected radically (according to the 8th edition of the International Association for lung cancer research (IASLC) breast cancer staging manual);
5. Patients with sufficient lung function;
6. Patients who need to obtain tumor tissue for EGFR mutation detection before operation, and no sensitive mutation was found in the EGFR detection results; 7. Patients with measurable target lesions according to the RECIST 1.1 standard;

8. Patients who have not received anti-tumor treatment for NSCLC; 9. Patients with normal function of main organs; 10. The fertile female patients must carry out the serum pregnancy test within 72 hours before the first medication, and the result is negative. The fertile female subjects and the male subjects whose partners are fertile females must agree to use efficient methods of contraception and lactation during the study period and within 90 days after the last administration of the study drug.

Exclusion Criteria:

1. Patients with tumor metastasis and known EGFR driving gene mutation;
2. Patients who have received any anti-tumor treatment in the past, including radiotherapy, chemotherapy, immunotherapy and anti-tumor treatment with traditional Chinese medicine;
3. Imaging (CT or MRI) shows that the tumor invades into the large blood vessels or the border with the blood vessels is unclear; or imaging (CT or MRI) shows that there is any pulmonary cavity or necrotic lesions;
4. Patients with any active autoimmune disease or history of autoimmune disease;
5. Patients with innate or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B, hepatitis C or co infection with hepatitis B and hepatitis C;
6. Patients with uncontrollable third cavity effusion, such as massive pleural effusion or ascites or pericardial effusion;
7. Routine urine test indicated that urine protein was >= (+ +), or 24-hour urine protein was >= 1g, or severe liver and kidney dysfunction;
8. Subjects requiring systemic treatment with corticosteroids (> 10 mg / day of prednisone or its equivalent) or other immunosuppressants within 14 days prior to the first administration;
9. Patients with other malignant tumors in the past 5 years;
10. Patients with previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiologic pneumonia, drug-induced pneumonia and active pneumonia confirmed by imaging;
11. Patients with uncontrollable hypertension (systolic blood pressure >= 140 mmHg or diastolic blood pressure >= 90 mmHg, despite the best drug treatment);
12. Patients with cardiac insufficiency;
13. Patients who have had arteriovenous thrombosis events within 6 months, such as cerebrovascular accident (including cerebral hemorrhage, cerebral infarction, transient ischemic attack, etc.);
14. Patients who underwent major surgery, open biopsy or significant trauma within 28 days before admission;
15. Patients with hemoptysis, active bleeding, ulcer, intestinal perforation and intestinal obstruction within 3 months before admission;
16. Patients who are taking part in other clinical studies or the time of the first medication is less than 4 weeks from the end of the previous clinical study (the last medication);
17. Patients with severe infection or fever of unknown origin > 38.5 degrees C within 4 weeks before medication;
18. Patients with known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
19. Pregnant or lactating women; those with fertility who are unwilling or unable to take effective contraceptive measures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) Rate | Up to 8weeks following completion of neoadjuvant treatment (up to Study Week 12)
  mPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) Rate | Up to 8weeks following completion of neoadjuvant treatment (up to Study Week 12)
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
Event Free Survival (EFS) | up to 5 years
  EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. EFS determined by biopsy assessed by investigator using RECIST 1.1 .
Objective Response (OR) | up to 6 weeks
  Objective response is defined as a complete response or partial response, as determined by the investigator according to RECIST v1.1
Disease-Free Survival (DFS) | up to 5 years
  DFS is defined as the time from the first date of no disease to local or distant recurrence or death due to any cause, whichever occurs first, as determined by the investigator during the adjuvant treatment and observation follow-up
Adverse Events (AEs) | up to 17 weeks
  The number of participants experiencing an AE will be assessed